CLINICAL TRIAL: NCT02311972
Title: Temperature Monitoring With InnerSense Esophageal Temperature Sensor/Feeding Tube After Birth Through Stabilization in VLBW Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Philips Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00051454
Record Dates: First submitted 2014-12-04; First posted 2014-12-09 (Estimated); Results first posted 2017-06-14 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-05

CONDITIONS: Body Temperature
MeSH Terms: interventions — Enteral Nutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control - Standard of Care (Active Comparator): Infants in the standard of care group will receive no study interventions other than study recorded axillary temperatures on admission, and at 1, 4, 8 and 24 hours. Infants will receive standard delivery room stabilization and NICU stabilization. Infants in the control group will receive a feeding tube as standard of care, and the standard issue feeding tube used in the Intensive Care Nursery does not have the capability to record or display esophageal temperatures. Nurses will record an axillary temperature upon admission to the NICU, and at 1, 4, 8 and 24 hours of age for each infant in both groups on a data sheet at the bedside. These data will be entered into a RedCap data base created for the study.
  Interventions: Device: Standard of care feeding tube
- Philips InnerSense Esophageal Temperature Sensor/Feeding Tube (Active Comparator): The nurse will insert an InnerSense temperature sensor/feeding tube per normal standards as soon after birth as possible, during delivery room stabilization. Nurses will record an axillary temperature upon admission to the NICU, and at 1, 4, 8 and 24 hours of age. The InnerSense tube will be attached to the infant's bedside monitor to continuously display esophageal temperatures. The tube will stay in place until the infant is 24 hours of age. Central body temperature will be displayed continuously for care-providers in the delivery room, through transport from the birthing center to the NICU and through stabilization. Infants will have a thermistor placed on the abdominal skin with standard skin tape once admitted in the NICU. This thermistor will be attached to a Squirrel SQ2010 (Grant Instruments) temperature monitor/data logger to collect abdominal temperatures every minute for the first 24 hours of life. All temperatures entered into the study database.
  Interventions: Device: Philips InnerSense Esophageal Temperature Sensor/Feeding Tube

INTERVENTIONS:
Device: Philips InnerSense Esophageal Temperature Sensor/Feeding Tube
  Arms: Philips InnerSense Esophageal Temperature Sensor/Feeding Tube
Device: Standard of care feeding tube
  Arms: Control - Standard of Care

SUMMARY:
Very low birth weight (VLBW) infants (<1500 grams at birth) and other low birth weight infants experience hypothermia after birth and through stabilization (first 24 hours of life) due to an inability to keep warm through metabolic heat production while experiencing heat loss during care.

The investigator hypothesizes that inserting an InnerSense oral gastric tube (Philips Healthcare) with its imbedded thermistor and attaching the tube to a temperature monitor with a digital temperature display will enable care-providers to monitor continuous body temperature and prompt them to provide warmth and prevent heat loss, thus preventing hypothermia in these infants for the first 24 hours of life. The investigator predicts infants in the intervention group will have warmer axillary temperatures upon admission to the NICU and at 1, 4, and 8 hours of age. Mothers in non-active labor will be sought for consent to enroll their VLBW infant into this study after the infant's birth. 160 VLBW infants and other low birth weight infants 1000-2000 grams will be randomized to the intervention group (placement of InnerSense oral gastric tube with thermistor to a Squirrel monitor for continuous digital temperature display, immediately after birth through 24 hours of life) or the control group (standard delivery room care and stabilization care). The study staff plans to enroll 180 infants (90 per group) to allow for screen failures. Axillary temperatures of all infants will be recorded at NICU admission, 1, 4, 8 and 24 hours of age. Further, the study staff intends to enroll approximately 300 Intensive Care Nursery providers who care for an InnerSense study infant and wish to complete a provider satisfaction survey. These providers will be asked to provide consent prior to completing the survey and their names will be recorded on a separate study enrollment log.

Infant demographic data will be compared to make sure groups are not significantly different. Temperatures from the intervention group will be compared to the control group using a student t test at each time point. Satisfaction questionnaires will be summarized and described. The InnerSense oral gastric tube with temperature monitoring is FDA approved for use and is being marketed commercially by Philips Healthcare. VLBW infants have oral gastric tubes placed as standard of care for feeding, and intermittently in the delivery room when positive pressure ventilation is necessary for respiratory stabilization. There are no additional safety risks to the intervention of this study; however, a safety/data monitoring committee will be formed and meet quarterly to monitor the trial.

ELIGIBILITY:
Inclusion Criteria:

* Parents of eligible infants must be enrolled prior to, or shortly after delivery as the InnerSense esophageal temperature sensor/feeding tube will be inserted post delivery resuscitation

Exclusion Criteria:

* Infants are excluded if parents were not consented prior to, or shortly after delivery
* Infants are not eligible if they have major congenital anomalies including gastrointestinal or facial abnormalities
* Infants with major cardiac anomalies are also excluded

Ages: 1 Minute to 24 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2014-11; Primary Completion 2016-04 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robin B Dail (Knobel), PhD, RN, FAAN, Principal Investigator — Duke University School of Nursing & School of Medicine, Department of Pediatrics
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Background] Martin JA, Hamilton BE, Ventura SJ, Osterman MJ, Mathews TJ. Births: final data for 2011. Natl Vital Stat Rep. 2013 Jun 28;62(1):1-69, 72. PMID 24974591
- [Background] Bhatt DR, White R, Martin G, Van Marter LJ, Finer N, Goldsmith JP, Ramos C, Kukreja S, Ramanathan R. Transitional hypothermia in preterm newborns. J Perinatol. 2007 Dec;27 Suppl 2:S45-7. doi: 10.1038/sj.jp.7211842. PMID 18034181
- [Background] Basu S, Rathore P, Bhatia BD. Predictors of mortality in very low birth weight neonates in India. Singapore Med J. 2008 Jul;49(7):556-60. PMID 18695864
- [Background] Laptook AR, Salhab W, Bhaskar B; Neonatal Research Network. Admission temperature of low birth weight infants: predictors and associated morbidities. Pediatrics. 2007 Mar;119(3):e643-9. doi: 10.1542/peds.2006-0943. Epub 2007 Feb 12. PMID 17296783
- [Background] Knobel RB, Wimmer JE Jr, Holbert D. Heat loss prevention for preterm infants in the delivery room. J Perinatol. 2005 May;25(5):304-8. doi: 10.1038/sj.jp.7211289. PMID 15861196
- [Background] Almeida PG, Chandley J, Davis J, Harrigan RC. Use of the heated gel mattress and its impact on admission temperature of very low birth-weight infants. Adv Neonatal Care. 2009 Feb;9(1):34-9. doi: 10.1097/01.ANC.0000346094.28110.11. PMID 19212164
- [Background] te Pas AB, Lopriore E, Dito I, Morley CJ, Walther FJ. Humidified and heated air during stabilization at birth improves temperature in preterm infants. Pediatrics. 2010 Jun;125(6):e1427-32. doi: 10.1542/peds.2009-2656. Epub 2010 May 10. PMID 20457686

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of 52 enrolled infants, 20 infants were randomized. Of those not randomized, 18 were over/underweight, 8 mothers were discharged prior to delivery/lost to contact, 5 infants were not enrolled due to no page at infant delivery and 1 was not enrolled because the infant did not a require feeding tube per attending physician at delivery.
Groups:
- Control - Standard of Care: Infants in the standard of care group will receive no study interventions other than study recorded axillary temperatures on NICU Admission, 1, 4, 8 and 24 hours of age. Infants will receive standard delivery room stabilization and NICU stabilization. Infants in the control group will receive a feeding tube as standard of care, and the standard issue feeding tube used in the Intensive Care Nursery does not have the capability to record or display esophageal temperatures.
- Philips InnerSense Esophageal Temperature Sensor/Feeding Tube: Infants will have an InnerSense temperature sensor/feeding tube inserted per normal standards as soon after birth as possible, during delivery room stabilization. Axillary temperature will be recorded upon NICU Admission, at 1, 4, 8 and 24 hours of age. The InnerSense tube will be attached to the infant's bedside monitor to continuously display esophageal temperatures. The tube will stay in place until the infant is 24 hours of age. Central body temperature will be displayed continuously for care-providers in the delivery room, through transport from the birthing center to the NICU and through stabilization. Infants will have a thermistor placed on the abdominal skin with standard skin tape once admitted in the NICU. This thermistor will be attached to a Squirrel SQ2010 (Grant Instruments) temperature monitor/data logger to collect abdominal temperatures every minute for the first 24 hours of life.
Period: Overall Study
Arm/Group | Control - Standard of Care | Philips InnerSense Esophageal Temperature Sensor/Feeding Tube
Started | 12 | 8
Completed | 12 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control - Standard of Care | Philips InnerSense Esophageal Temperature Sensor/Feeding Tube | Total
Number analyzed (Participants) | 12 | 8 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 12 | 8 | 20
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 5 | 14
  Male | 3 | 3 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 12 | 6 | 18
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 8 | 20

OUTCOME MEASURES:

1. Primary Outcome: Mean Axillary Admission Temperature
Description: Mean axillary temperatures upon Admission from infants in the InnerSense group and the standard of care group will be compared to determine if a significant difference
Time Frame: Admission
Measure: Mean (Standard Deviation); unit: Degrees Celsius
Arm/Group | Control - Standard of Care | Philips InnerSense Esophageal Temperature Sensor/Feeding Tube
Number analyzed (Participants) | 12 | 8
Degrees Celsius | 36.77 (0.61) | 36.68 (0.51)
Statistical Analysis 1: Comparison: Control - Standard of Care vs Philips InnerSense Esophageal Temperature Sensor/Feeding Tube; Test type: Superiority — Mean axillary admission temperature; p = 0.7294, t-test, 2 sided

2. Primary Outcome: Mean Axillary Temperature at 4 Hours of Infant Life
Description: The mean axillary temperature at 4 hours of age will be compared for infants in the InnerSense group and the standard of care group to determine if a significant difference is seen at 4 hours of life.
Time Frame: 4 Hours of Infant Life
Measure: Mean (Standard Deviation); unit: Degrees Celsius
Arm/Group | Control - Standard of Care | Philips InnerSense Esophageal Temperature Sensor/Feeding Tube
Number analyzed (Participants) | 12 | 8
Degrees Celsius | 36.93 (0.27) | 36.74 (0.42)
Statistical Analysis 1: Comparison: Control - Standard of Care vs Philips InnerSense Esophageal Temperature Sensor/Feeding Tube; Test type: Superiority; p = 0.2360, t-test, 2 sided

3. Secondary Outcome: Percentage of Infants With Hypothermic Temperatures (<36.5° C) Upon Admission
Description: Axillary temperatures for infants in the InnerSense group and infants in the standard of care group will be compared on admission to determine the percentage of hypothermia in both groups.
Time Frame: Admission
Measure: Count of Participants; unit: Participants
Arm/Group | Control - Standard of Care | Philips InnerSense Esophageal Temperature Sensor/Feeding Tube
Number analyzed (Participants) | 12 | 8
Participants | 5 | 3
Statistical Analysis 1: Comparison: Control - Standard of Care vs Philips InnerSense Esophageal Temperature Sensor/Feeding Tube; Test type: Superiority; p = 0.05, t-test, 2 sided

4. Secondary Outcome: Percentage of Infants With Hypothermic Temperatures (<36.5° C) at 1 Hour of Infant Life
Description: Axillary temperatures for infants in the InnerSense group and infants in the standard of care group will be compared at 1 hour to determine the percentage of hypothermia in both groups.
Time Frame: 1 Hour of Infant Life
Measure: Count of Participants; unit: Participants
Arm/Group | Control - Standard of Care | Philips InnerSense Esophageal Temperature Sensor/Feeding Tube
Number analyzed (Participants) | 12 | 8
Participants | 1 | 4
Statistical Analysis 1: Comparison: Control - Standard of Care vs Philips InnerSense Esophageal Temperature Sensor/Feeding Tube; Test type: Superiority; p = 0.1089, t-test, 2 sided

5. Secondary Outcome: Percentage of Infants With Hypothermic Temperatures (<36.5° C) at 4 Hours of Infant Life
Description: Axillary temperatures for infants in the InnerSense group and infants in the standard of care group will be compared at 4 hours to determine the percentage of hypothermia in both groups.
Time Frame: 4 Hours of Infant Life
Measure: Count of Participants; unit: Participants
Arm/Group | Control - Standard of Care | Philips InnerSense Esophageal Temperature Sensor/Feeding Tube
Number analyzed (Participants) | 12 | 8
Participants | 1 | 1
Statistical Analysis 1: Comparison: Control - Standard of Care vs Philips InnerSense Esophageal Temperature Sensor/Feeding Tube; Test type: Superiority; p = 0.05, t-test, 2 sided

6. Secondary Outcome: Percentage of Infants With Hypothermic Temperatures (<36.5° C) at 8 Hours of Infant Life
Description: Axillary temperatures for infants in the InnerSense group and infants in the standard of care group will be compared at 8 hours to determine the percentage of hypothermia in both groups.
Time Frame: 8 Hours of Infant Life
Measure: Count of Participants; unit: Participants
Arm/Group | Control - Standard of Care | Philips InnerSense Esophageal Temperature Sensor/Feeding Tube
Number analyzed (Participants) | 12 | 8
Participants | 2 | 0
Statistical Analysis 1: Comparison: Control - Standard of Care vs Philips InnerSense Esophageal Temperature Sensor/Feeding Tube; Test type: Superiority; p = 0.4947, t-test, 2 sided

7. Secondary Outcome: Pearson Correlation Coefficient Comparing Thermistor Abdominal Temperature to Esophageal Temperature in Each Infant in the Experimental Arm.
Description: Temperatures measured by the abdomen thermistor will be compared with esophageal temperatures in each infant over 24 hours using pearson correlation coefficient.
Time Frame: Admission to 24 hours of infant life.
Population: Intervention Group Only: Two infants with the InnerSense did not have skin temperatures dowloaded from the data logger due to data logger malfunction and one infant had a Squirrel monitor attached to the InnerSense tube that did not read or log temperatures. Therefore only data from 5 infants was available to analyze.
Measure: Number; unit: Pearson Correlation Coefficient
Groups:
- Philips InnerSense Esophageal Temperature Sensor/Feeding Tube: The nurse will insert an InnerSense temperature sensor/feeding tube per normal standards as soon after birth as possible, during delivery room stabilization. Nurses will record an axillary temperature upon admission to the NICU, at 1, 4, 8 and 24 hours of age. The InnerSense tube will be attached to the infant's bedside monitor to continuously display esophageal temperatures. The tube will stay in place until the infant is 24 hours of age. Central body temperature will be displayed continuously for care-providers in the delivery room, through transport from the birthing center to the NICU and through stabilization. Infants will have a thermistor placed on the abdominal skin with standard skin tape once admitted in the NICU. This thermistor will be attached to a Squirrel SQ2010 (Grant Instruments) temperature monitor/data logger to collect abdominal temperatures every minute for the first 24 hours of life.
Arm/Group | Philips InnerSense Esophageal Temperature Sensor/Feeding Tube
Number analyzed (Participants) | 5
Pearson Correlation Coefficient
  Infant 007: number analyzed (Participants) | 1
  Infant 007 | 0.534
  Infant 010: number analyzed (Participants) | 1
  Infant 010 | 0.692
  Infant 015: number analyzed (Participants) | 1
  Infant 015 | 0.713
  Infant 039: number analyzed (Participants) | 1
  Infant 039 | 0.152
  Infant 040: number analyzed (Participants) | 1
  Infant 040 | 0.023
Statistical Analysis 1: Comparison: Philips InnerSense Esophageal Temperature Sensor/Feeding Tube; Test type: Superiority — Infant 007; p < 0.0001, t-test, 2 sided
Statistical Analysis 2: Comparison: Philips InnerSense Esophageal Temperature Sensor/Feeding Tube; Test type: Superiority — Infant 010; p < 0.0001, t-test, 2 sided
Statistical Analysis 3: Comparison: Philips InnerSense Esophageal Temperature Sensor/Feeding Tube; Test type: Superiority — Infant 015; p < 0.0001, t-test, 2 sided
Statistical Analysis 4: Comparison: Philips InnerSense Esophageal Temperature Sensor/Feeding Tube; Test type: Superiority — Infant 039; p < 0.0001, t-test, 2 sided
Statistical Analysis 5: Comparison: Philips InnerSense Esophageal Temperature Sensor/Feeding Tube; Test type: Superiority — Infant 040; p = 0.3947, t-test, 2 sided

8. Other Pre Specified Outcome: Exploratory Outcome: Caregiver Satisfaction and Ease of Use
Description: Describe the caregiver satisfaction and ease of use for the InnerSense by using a provider questionnaire. Caregivers will rate the InnerSense feeding tube with traditional feeding tubes used in the Intensive Care Nursery.
Time Frame: First 24 hours of infant life.
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from time of randomization to study completion, approximately 24 hours.
Description: Adverse events were defined as any harm suffered by the infant related to the study procedures or instruments or a death of an infant while under study protocol. An adverse event was determined if the infants decompensation or bodily injury was related to the study procedures.
Arm/Group | Control - Standard of Care | Philips InnerSense Esophageal Temperature Sensor/Feeding Tube
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/8
Other Adverse Events (participants affected / at risk) | 0/12 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No